CLINICAL TRIAL: NCT01775839
Title: Clinical Trial to Evaluate the Influence of Genotype of Drug Metabolizing Enzyme or Transporter and Drug-drug Interactions of Aspirin Co-administration on the PK/PD of Clopidogrel and PK of Digoxin in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate the Influence of Genotype and DDIs of Aspirin on the PK/PD of Clopidogrel and PK of Digoxin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PGX_Clopidogrel_002
Record Dates: First submitted 2013-01-15; First posted 2013-01-25 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: DRUG REACTIONS
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Aspirin; Clopidogrel; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin+Clopidogrel/Digoxin(oral) (Experimental): Aspirin: Day 1 ~ Day 59(~65; till the EGC) Clopidogrel: Day -3, 26, 54 Digoxin: Day -2, 27, 55
  Interventions: Drug: Aspirin+Clopidogrel/Digoxin(oral)
- Aspirin+Clopidogrel/Digoxin(IV) (Experimental): Aspirin: Day 1 ~ Day 59(~65; till the EGC) Clopidogrel: Day -3, 26, 54 Digoxin: Day -2, 27, 55
  Interventions: Drug: Aspirin+Clopidogrel/Digoxin(IV)

INTERVENTIONS:
Drug: Aspirin+Clopidogrel/Digoxin(oral) — oral administration of digoxin
  Other Names: Aspirin; Clopidogrel; Digoxin
  Arms: Aspirin+Clopidogrel/Digoxin(oral)
Drug: Aspirin+Clopidogrel/Digoxin(IV) — intravenous administration of digoxin
  Other Names: Aspirin; Clopidogrel; Digoxin
  Arms: Aspirin+Clopidogrel/Digoxin(IV)

SUMMARY:
Clinical trial to evaluate the influence of multiple aspirin administration on PK and PD of co-administered drugs

DETAILED DESCRIPTION:
Clinical trial to evaluate the influence of genotype of drug metabolizing enzyme or transporter and drug-drug interactions of aspirin co-administration on the pharmacokinetics / pharmacodynamics of clopidogrel and pharmacokinetics of digoxin in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years.
* A body weight in the range of 50 kg (inclusive) - 90 kg (exclusive) and a body mass index (BMI) in the range 18.5 kg/m2 (inclusive) - 27 kg/m2 (inclusive).
* Sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully. informed about the study procedures.

Exclusion Criteria:

* Presence or history of hypersensitivity or allergic reactions to drugs including investigational product (clopidogrel, digoxin or aspirin)
* Clinically relevant abnormal medical history that could interfere with the objectives of the study.
* A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug.
* A subject whose lab test results are as follows; Platelet count or PT, aPTT < 0.9 x lower limit of reference range of > 1.1 x upper limit of reference range.
* A subject whose SBP is over 160 mmHg or below 90 mmHg and DBP is over 100 mmHg or below 50 mmHg.
* Clinically significant abnormal findings of ECG during screening test.
* Presence or history of drug abuse or positive result in urine drug screening test.
* Participation in other clinical trial within 2 months before first dose.
* Use of CYP inducer (ex. rifampin) within 4 weeks before first dose.
* Use of a prescription medicine, herbal medicine within 2 weeks or over-the-counter medication or vitamin substances within 1 week before first dose.
* Use of grapefruit juice within 1 week before first dose.
* Blood donation during 2 months or apheresis during 1 month before the study.
* Use of alcohol over 21 units/weeks
* Smoking of more than 10 cigarettes/days within 3 months before first dose.
* Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
AUC and Cmax of Clopidogrel and Digoxin | pre- and post dose of Clopidogrel, Digoxin administration
  (Clopidogrel)Predose and 10, 20, 30, 40, 50 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 h postdose on Week 0, 4, 8 (Digoxin) Predose and 10, 20, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 h postdose on Week 0, 4, 8

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, Principal Investigator — SNUH
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea